CLINICAL TRIAL: NCT06118827
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Doses of HS-10518 in Healthy Adult Premenopausal Females in China
Brief Title: A Study of HS-10518 in Healthy Female Participants
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HS-10518-101
Record Dates: First submitted 2023-10-24; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — TU2670

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- HS-10518 Dose 1 (Experimental): Dose level 1 of HS-10518, QD, orally, 7 days
  Interventions: Drug: HS-10518
- Placebo Dose 1 (Placebo Comparator): Dose level 1 of matching placebo, QD, orally, 7 days
  Interventions: Drug: Placebo
- HS-10518 Dose 2 (Experimental): Dose level 2 of HS-10518, QD, orally, 7 days
  Interventions: Drug: HS-10518
- Placebo Dose 2 (Placebo Comparator): Dose level 2 of matching placebo, QD, orally, 7 days
  Interventions: Drug: Placebo
- HS-10518 Dose 3 (Experimental): Dose level 3 of HS-10518, QD, orally, 7 days
  Interventions: Drug: HS-10518
- Placebo Dose 3 (Placebo Comparator): Dose level 3 of matching placebo,QD, orally, 7 days
  Interventions: Drug: Placebo
- HS-10518 Dose 4 (Experimental): Dose level 4 of HS-10518, QD, orally, 7 days
  Interventions: Drug: HS-10518
- Placebo Dose 4 (Placebo Comparator): Dose level 4 of matching placebo, QD, orally, 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HS-10518 — QD, orally for 7 days
  Other Names: TU2670
  Arms: HS-10518 Dose 1; HS-10518 Dose 2; HS-10518 Dose 3; HS-10518 Dose 4
Drug: Placebo — QD, orally for 7 days
  Other Names: HS-10518 Placebo
  Arms: Placebo Dose 1; Placebo Dose 2; Placebo Dose 3; Placebo Dose 4

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of HS-10518 in healthy adult premenopausal females in China.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, multiple-dose, single-center phase 1 study in Chinese healthy premenopausal females aged 18-45 years with a regular menstrual cycle (26-32 days). The main purpose of the study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of HS-10518, a gonadotropin-releasing hormone antagonist.

About 48 eligible female subjects will be enrolled. The study contains four cohorts.

In each cohort, participants will be randomly assigned to the HS-10518 arm or the placebo arm in a 3:1 ratio. HS-10518/matching placebo will be administered from Day 1 to Day 7. The study duration of each participant is up to ~10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* • Subject is a healthy premenopausal female aged 18-45 (inclusive) at Screening;

  * Subject has a body weight ≥45kg with a body mass index (BMI) of 18-28 kg/m^2 (inclusive);
  * Subject has a normal menstrual cycle for no less than 2 years (Cycle: 26-32 days, menstrual period: 2-7 days), and have a positive ovulation test in the cycle prior to drug administration;
  * Subject is willing to use highly effective, non-hormone contraceptive methods from signing the consent form until 3 months after the last dose;
  * Subject agrees to draw blood in pre-specified time points throughout the study and to attend the follow-up visit;
  * Subject is able to understand the purpose, process and potential adverse events of the study, and is willing to sign a written informed consent form.

Exclusion Criteria:

* • Subject took caffeine-rich or xanthine-rich food or drink (e.g. coffee, tea, chocolate, cola, etc.), tobacco or alcoholic products within 48 hours prior to drug administration;

  * Subject took any grapefruit, grapefruit juice or other products within 7 days prior to first dose of study drug;
  * Subject has a positive breath alcohol test or a history of alcohol abuse;
  * Subject is a heavy smoker, or smokes ≥5 cigarettes per day, or is not able to cease smoking during the study (including e-cigarette);
  * Subject has a history of drug abuse or a positive urine drug test;
  * Subject is pregnant, breastfeeding or has a positive pregnancy test at Screening

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AE) as assessed by CTCAE v4.0 | From screening to day 16
  Assessment of safety and tolerability of multiple-dose HS-10518 in healthy female subjects in terms of the frequency, severity and causality of AEs, serious adverse events (SAEs) and AEs leading to study discontinuation. CTCAE v4.0 will be used for classification and severity determination.
Assessment of safety and tolerability of HS-10518 in terms of the frequency, severity and causality of AEs, serious adverse events (SAEs) and AEs leading to study discontinuation. | From screening to day 16
  Incidence of any markedly abnormal standard vital sign measurements is collected throughout study.
Incidence of clinically significant abnormal findings in 12-lead electrocardiogram (ECG) | From screening to day 16
  Incidence of any clinically significant abnormal findings in 12-lead ECG is collected throughout study.

SECONDARY OUTCOMES:
Plasma pharmacokinetic (PK) parameter: Maximum plasma concentration (Cmax) | Day 1 (after the first dose) and Day 7-10 (after the last dose)
  The maximum observed plasma concentration of HS-10518.
PK parameter :Time of maximum observed plasma concentration (Tmax) | Day 1 (after the first dose) and Day 7-10 (after the last dose)
  Time of the maximum observed plasma concentration of HS-10518.
PK parameter: Area under the concentration-time curve from time 0 to the last quantifiable concentration (AUC0-t) | Day 1 (after the first dose) and Day 7-10 (after the last dose)
  Area under the concentration-time curve from time 0 to the last quantifiable concentration of HS-10518.